CLINICAL TRIAL: NCT01214889
Title: Immunogenicity and Safety of the Sanofi Pasteur's DTacP-IPV//PRP~T Combined Vaccine (PENTAXIM™) Versus Sanofi Pasteur's DTacP-IPV Combined Vaccine (TETRAXIM™) Given Simultaneously at Separate Sites With PRP~T Conjugate Vaccine (ACTHIB™) as a Three-dose Primary Vaccination at 2, 4 and 6 Months of Age in South Korean Infants
Brief Title: Study of PENTAXIM™ Vaccine Versus TETRAXIM™ Vaccine Given With ACTHIB™ Vaccine in South Korean Infants.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E2I49; U1111-1115-6381 (Other: WHO)
Record Dates: First submitted 2010-10-01; First posted 2010-10-05 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Diphtheria; Tetanus; Pertussis; Poliomyelitis; Haemophilus Influenzae Type B
Keywords: Diphtheria; Tetanus; Pertussis; Haemophilus influenzae type B; Poliomyelitis; PENTAXIM™; TETRAXIM™
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis; Haemophilus Infections | interventions — Pentavac; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group A (Experimental): Participants will receive a single dose of DTacP-IPV//PRP T combined vaccine (PENTAXIM™) at age 2, 4 and 6 months.
  Interventions: Biological: PENTAXIM™: DTacP IPV//PRP~T combined vaccine
- Study Group B (Active Comparator): Participants will receive a dose of DTacP IPV combined vaccine (TETRAXIM™) and PRP-T vaccine (ActHIB™) at 2, 4, and 6 months of age.
  Interventions: Biological: TETRAXIM™: DTacP IPV combined vaccine and ActHIB™: PRP tetanus conjugate vaccine

INTERVENTIONS:
Biological: PENTAXIM™: DTacP IPV//PRP~T combined vaccine — 0.5 mL, intramuscular
  Other Names: PENTAXIM™
  Arms: Study Group A
Biological: TETRAXIM™: DTacP IPV combined vaccine and ActHIB™: PRP tetanus conjugate vaccine — 0.5 mL of each vaccine; intramuscular
  Other Names: TETRAXIM™; ActHIB™
  Arms: Study Group B

SUMMARY:
This study is designed to assess the immunogenicity and safety of PENTAXIM™ combined vaccine versus TETRAXIM™ vaccine to support registration of PENTAXIM™ in South Korea.

Primary Objective:

To demonstrate the non-inferiority in terms of seroprotection rates (Diphtheria, Tetanus, Polio types 1, 2 and 3, Polyribosyl Ribitol Phosphate [PRP]) and vaccine response rates to acellular Pertussis antigens of sanofi pasteur's PENTAXIM™ vaccine versus sanofi pasteur's TETRAXIM™ and Act (Haemophilus influenzae type b) HIB™ vaccines, one month after the three-dose primary vaccination.

DETAILED DESCRIPTION:
All participants will receive three primary doses of their assigned study the vaccine, on Days 0, 60, and 120. They will be assessed for immunogenicity on Day 0 before vaccination and Day 150 post-vaccination. Safety will be assessed for all participants throughout the study, up to Day 157.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 months (56 to 70 days) inclusive on the day of inclusion
* Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg
* Informed consent form signed by the parent(s) or other legal representative
* Able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the trial inclusion
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as long term systemic corticosteroids therapy
* Systemic hypersensitivity to any of the vaccine components or history of a life threatening reaction to the trial vaccine or a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion
* Blood or blood derived products received in the past or current or planned administration during the trial (including immunoglobulins).
* Any vaccination in the 3 weeks preceding the first trial vaccination.
* History of diphtheria, tetanus, pertussis, poliomyelitis, Haemophilus influenzae type b infection (confirmed either clinically, serologically or microbiologically).
* Clinical or known serological evidence of systemic illness including Hepatitis B, Hepatitis C and/or Human Immunodeficiency Virus (HIV) infection
* Previous vaccination against the diphtheria, tetanus, pertussis, poliomyelitis diseases or Haemophilus influenzae type b infection with the trial vaccine or another vaccine.
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
* History of/current major neurological diseases or seizures.
* Febrile illness (axillary temperature ≥ 38ºC) or acute illness on the day of inclusion.
* Known family history of congenital or genetic immuno-deficiency.

Ages: 56 Days to 70 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 370 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Non-inferiority in terms of seroprotection rates (Diphtheria, Tetanus, Polio types 1, 2 and 3, Polyribosyl Ribitol Phosphate conjugated to Tetanus protein) of PENTAXIM™ Vaccine to the Tetraxim™ and PRP~T conjugate (Act-HIB™) vaccines. | 1 month post-dose 3 vaccination

SECONDARY OUTCOMES:
Information regarding the safety (in terms of solicited injection site and systemic reactions) of PENTAXIM™ vaccine. | Day 0 up to Day 157

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (5):
- South Korea (5):
  - Daejeon
  - Gyeionggi Do
  - Gyeonggi-do
  - Incheon
  - Seoul

REFERENCES:
- [Derived] Kang JH, Lee HJ, Kim KH, Oh SH, Cha SH, Lee J, Kim NH, Eun BW, Kim CH, Hong YJ, Kim HH, Lee KY, Kim YJ, Cho EY, Kim HS, Guitton F, Ortiz E. The Immunogenicity and Safety of a Combined DTaP-IPV//Hib Vaccine Compared with Individual DTaP-IPV and Hib (PRP~T) Vaccines: a Randomized Clinical Trial in South Korean Infants. J Korean Med Sci. 2016 Sep;31(9):1383-91. doi: 10.3346/jkms.2016.31.9.1383. PMID 27510380
- See also: Related Info — http://www.sanofipasteur.com